CLINICAL TRIAL: NCT02106923
Title: Relative Bioavailability of Two Newly Developed FDC Tablet Strengths (10 mg/1000 mg and 5mg/750mg) of Empagliflozin/Metformin Extended Release Compared With the Free Combination of Empagliflozin and Metformin Extended Release in Healthy Subjects (an Open-label, Randomised, Single Dose, Two-way Crossover Study)
Brief Title: Relative Bioavailability of 2 Fixed Dose Combinations of Empagliflozin/Metformin Extended Release (XR) Compared With Single Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.14
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Healthy

ARMS (3):
- High dose, fasted (Experimental): 1 fixed dose combination (FDC) tablet vs 3 single tablets under fasted conditions
  Interventions: Drug: 10 mg Empagliflozin/1000 mg Metformin XR; Drug: 1 tablet Empagliflozin/2 tablets Metformin XR
- High dose, fed (Experimental): 1 fixed dose combination (FDC) tablet vs 3 single tablets under fed conditions
  Interventions: Drug: 1 tablet Empagliflozin/2 tablets Metformin XR; Drug: 10 mg Empagliflozin/1000 mg Metformin XR
- Low dose, fasted (Experimental): 2 fixed dose combination (FDC) tablets vs 4 single tablets under fasted conditions
  Interventions: Drug: 1 tablet 10 mg Empagliflozin/3 tablets Metformin XR; Drug: 2 tablets 5 mg Empagliflozin/750 Metformin XR

INTERVENTIONS:
Drug: 1 tablet Empagliflozin/2 tablets Metformin XR — Active Comparator: 1 x Empagliflozin/2x Metformin XR tablets
  Arms: High dose, fed
Drug: 10 mg Empagliflozin/1000 mg Metformin XR — Experimental: high dose Empagliflozin/Metformin XR, FDC tablet
  Arms: High dose, fasted
Drug: 1 tablet 10 mg Empagliflozin/3 tablets Metformin XR — Active Comparator: 1 x Empagliflozin/3 x Metformin XR tablets
  Arms: Low dose, fasted
Drug: 2 tablets 5 mg Empagliflozin/750 Metformin XR — Experimental:2 x low dose Empagliflozin/Metformin XR FDC tablets
  Arms: Low dose, fasted
Drug: 1 tablet Empagliflozin/2 tablets Metformin XR — Active Comparator: 1 x Empagliflozin/2x Metformin XR tablets
  Arms: High dose, fasted
Drug: 10 mg Empagliflozin/1000 mg Metformin XR — Experimental: high dose Empagliflozin/Metformin XR, FDC tablet
  Arms: High dose, fed

SUMMARY:
The purpose of this trial is to demonstrate the relative bioavailability of 2 newly developed fixed dose combinations (FDC) tablets containing empagliflozin & metformin XR and the single tablets of empagliflozin and metformin XR when administered singularly

ELIGIBILITY:
Inclusion criteria:

1. Healthy males or females
2. Age 18-50 years (incl.)
3. Body Mass Index (BMI) 18.5 to 29.9 kg/m2 (incl.)
4. Subjects must be able to understand and comply with study requirements

Exclusion criteria:

Any deviation from healthy condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Empa+1000mg Met FDC / Empa+1000mg Glumetza® (Fasted): Oral administration of 1 x 10 mg Empagliflozin (Empa)/1000 mg metformin (Met) extended release (XR) fixed dose combination (FDC) followed by oral administration of 1 x 10 mg Empagliflozin + 2 x 500 mg Glumetza® XR. Both treatments were taken with 240 mL of water after an overnight fast of at least 10 hours (h).
- Empa+1000mg Glumetza / Empa+1000mg Met FDC (Fasted): Oral administration of 1 x 10 mg Empagliflozin + 2 x 500 mg Glumetza® XR followed by oral administration of 1 x 10 mg Empagliflozin/1000 mg metformin XR FDC. Both treatments were taken with 240 mL of water after an overnight fast of at least 10 h.
- Empa+1000mg Met FDC / Empa+1000mg Glumetza (Fed): Oral administration of 1 x 10 mg Empagliflozin/1000 mg Metformin XR FDC followed by oral administration of 1 x 10 mg Empagliflozin + 2 x 500 mg Glumetza® XR. Both treatments were taken with 240 mL of water after a high-fat, high-caloric meal.
- Empa+1000mg Glumetza / Empa+1000mg Met FDC (Fed): Oral administration of 1 x 10 mg Empagliflozin + 2 x 500 mg Glumetza® XR followed by oral administration of 1 x 10 mg Empagliflozin/1000 mg Metformin XR FDC. Both treatments were taken with 240 mL of water after a high-fat, high-caloric meal.
- Empa+1500mg Met FDC / Empa+1500mg Glumetza (Fasted): Oral administration of 2 x 5 mg Empagliflozin/750 mg Metformin XR FDC followed by oral administration of 1 x 10 mg Empagliflozin + 3 x 500 mg Glumetza® XR. Both treatments were taken with 240 mL of water after an overnight fast of at least 10 h.
- Empa+1500mg Glumetza / Empa+1500mg Met FDC (Fasted): Oral administration of 1 x 10 mg Empagliflozin + 3 x 500 mg Glumetza® XR followed by oral administration of 2 x 5 mg Empagliflozin/750 mg Metformin XR FDC. Both treatments were taken with 240 mL of water after an overnight fast of at least 10 h.
Period: Overall Study
Arm/Group | Empa+1000mg Met FDC / Empa+1000mg Glumetza® (Fasted) | Empa+1000mg Glumetza / Empa+1000mg Met FDC (Fasted) | Empa+1000mg Met FDC / Empa+1000mg Glumetza (Fed) | Empa+1000mg Glumetza / Empa+1000mg Met FDC (Fed) | Empa+1500mg Met FDC / Empa+1500mg Glumetza (Fasted) | Empa+1500mg Glumetza / Empa+1500mg Met FDC (Fasted)
Started | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set which included all subjects who were dispensed study medication and were documented to have taken at least one dose of study drug.
Groups:
- 1000mg, Fasted: Patients orally administered either 1 x 10 mg Empagliflozin/1000 mg metformin (Met) XR FDC or 1 x 10 mg Empagliflozin + 2 x 500 mg Glumetza® XR. Both treatments were taken with 240 mL of water after an overnight fast of at least 10 hours (h).
- 1000mg, Fed: Patients orally administered either 1 x 10 mg Empagliflozin/1000 mg Metformin XR FDC or 1 x 10 mg Empagliflozin + 2 x 500 mg Glumetza® XR. Both treatments were taken with 240 mL of water after a high-fat, high-caloric meal
- 1500mg, Fasted: Patients orally administered either 2 x 5 mg Empagliflozin/750 mg Metformin XR FDC or 1 x 10 mg Empagliflozin + 3 x 500 mg Glumetza® XR. Both treatments were taken with 240 mL of water after an overnight fast of at least 10 h
- Total: Total of all reporting groups
Arm/Group | 1000mg, Fasted | 1000mg, Fed | 1500mg, Fasted | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (8.7) | 32.4 (9.1) | 31.3 (8.7) | 30.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 16 | 48
  Male | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point), for Empagliflozin
Description: Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h, 1h 20min, 1h 40min, 2h, 2.5h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h, 16h, 24h, 36h, 48h and 72h after drug administration
Population: Pharmacokinetic (PK) set (PKS) which included all subjects of the treated set who provided at least one observation for at least one primary PK endpoint and had no important protocol violations with respect to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa/1000 mg Glumetza® (Fasted): Oral administration of 1 x 10 mg Empagliflozin + 2 x 500 mg Glumetza® XR with 240 mL of water after an overnight fast of at least 10 h
- Empa/ 1000 mg Met FDC (Fasted): Oral administration of 1 x 10 mg Empagliflozin/1000 mg metformin XR fixed dose combination (FDC) with 240 mL of water after an overnight fast of at least 10 h
- Empa/1000 mg Glumetza ® (Fed): Oral administration of 1 x 10 mg Empagliflozin + 2 x 500 mg Glumetza® XR with 240 mL of water after a high-fat, high-caloric meal
- Empa/ 1000 mg Met FDC (Fed): Oral administration of 1 x 10 mg Empagliflozin/1000 mg Metformin XR FDC with 240 mL of water after a high-fat, high-caloric meal
- Empa/ 1500 mg Glumetza® (Fasted): Oral administration of 1 x 10 mg Empagliflozin + 3 x 500 mg Glumetza® XR with 240 mL of water after an overnight fast of at least 10 h
- Empa/ 1500 mg Met FDC (Fasted): Oral administration of 2 x 5 mg Empagliflozin/750 mg Metformin XR FDC with 240 mL of water after an overnight fast of at least 10 h
Arm/Group | Empa/1000 mg Glumetza® (Fasted) | Empa/ 1000 mg Met FDC (Fasted) | Empa/1000 mg Glumetza ® (Fed) | Empa/ 1000 mg Met FDC (Fed) | Empa/ 1500 mg Glumetza® (Fasted) | Empa/ 1500 mg Met FDC (Fasted)
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 24 | 23
nmol*h/L | 2630 (18.9) | 2710 (18.3) | 2720 (20.5) | 2710 (19.9) | 2790 (17.3) | 2680 (18.7)
Statistical Analysis 1: Comparison: Empa/1000 mg Glumetza® (Fasted) vs Empa/ 1000 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 102.98, 90% CI 2-sided [100.505 to 105.514], Standard Error of Mean 1.014 — Ratio calculated as Empa/ 1000 mg Met FDC (Fasted) divided by Empa/1000 mg Glumetza® (Fasted)
Statistical Analysis 2: Comparison: Empa/1000 mg Glumetza ® (Fed) vs Empa/ 1000 mg Met FDC (Fed); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 100.25, 90% CI 2-sided [96.809 to 103.823], Standard Error of Mean 1.021 — Ratio calculated as Empa/ 1000 mg Met FDC (Fed) divided by Empa/1000 mg Glumetza ® (Fed)
Statistical Analysis 3: Comparison: Empa/ 1500 mg Glumetza® (Fasted) vs Empa/ 1500 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 96.08, 90% CI 2-sided [93.507 to 98.721], Standard Error of Mean 1.016 — Ratio calculated as Empa/ 1500 mg Met FDC (Fasted) divided by Empa/ 1500 mg Glumetza® (Fasted)

2. Primary Outcome: AUC0-tz (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point) for Metformin
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 to the last quantifiable data point
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Empa/1000 mg Glumetza® (Fasted) | Empa/ 1000 mg Met FDC (Fasted) | Empa/1000 mg Glumetza ® (Fed) | Empa/ 1000 mg Met FDC (Fed) | Empa/ 1500 mg Glumetza® (Fasted) | Empa/ 1500 mg Met FDC (Fasted)
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 24 | 23
ng*h/mL | 7020 (35.2) | 7170 (36.2) | 13500 (19.1) | 13200 (18.8) | 9860 (26.4) | 10100 (25.6)
Statistical Analysis 1: Comparison: Empa/1000 mg Glumetza® (Fasted) vs Empa/ 1000 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p = 0.0011, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 102.04, 90% CI 2-sided [92.30 to 112.81], Standard Error of Mean 1.06 — Ratio calculated as Empa/ 1000 mg Met FDC (Fasted) divided by Empa/1000 mg Glumetza® (Fasted)
Statistical Analysis 2: Comparison: Empa/1000 mg Glumetza ® (Fed) vs Empa/ 1000 mg Met FDC (Fed); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 98.93, 90% CI 2-sided [95.45 to 102.53], Standard Error of Mean 1.02 — Ratio calculated as Empa/ 1000 mg Met FDC (Fed) divided by Empa/1000 mg Glumetza ® (Fed)
Statistical Analysis 3: Comparison: Empa/ 1500 mg Glumetza® (Fasted) vs Empa/ 1500 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p = 0.0002, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 101.70, 90% CI 2-sided [93.59 to 110.52], Standard Error of Mean 1.05 — Ratio calculated as Empa/ 1500 mg Met FDC (Fasted) divided by Empa/ 1500 mg Glumetza® (Fasted)

3. Secondary Outcome: AUC0-infinity (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity), for Empagliflozin
Description: Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa/1000 mg Glumetza® (Fasted) | Empa/ 1000 mg Met FDC (Fasted) | Empa/1000 mg Glumetza ® (Fed) | Empa/ 1000 mg Met FDC (Fed) | Empa/ 1500 mg Glumetza® (Fasted) | Empa/ 1500 mg Met FDC (Fasted)
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 24 | 23
nmol*h/L | 2680 (18.7) | 2760 (17.9) | 2790 (21.3) | 2770 (20.2) | 2840 (17.4) | 2740 (19.5)
Statistical Analysis 1: Comparison: Empa/1000 mg Glumetza® (Fasted) vs Empa/ 1000 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 102.88, 90% CI 2-sided [100.446 to 105.373], Standard Error of Mean 1.014 — Ratio calculated as Empa/ 1000 mg Met FDC (Fasted) divided by Empa/1000 mg Glumetza® (Fasted)
Statistical Analysis 2: Comparison: Empa/1000 mg Glumetza ® (Fed) vs Empa/ 1000 mg Met FDC (Fed); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 100.03, 90% CI 2-sided [96.448 to 103.738], Standard Error of Mean 1.021 — Ratio calculated as Empa/ 1000 mg Met FDC (Fed) divided by Empa/1000 mg Glumetza ® (Fed)
Statistical Analysis 3: Comparison: Empa/ 1500 mg Glumetza® (Fasted) vs Empa/ 1500 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 96.49, 90% CI 2-sided [93.758 to 99.311], Standard Error of Mean 1.017 — Ratio calculated as Empa/ 1500 mg Met FDC (Fasted) divided by Empa/ 1500 mg Glumetza® (Fasted)

4. Primary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma, for Empagliflozin
Description: Maximum measured concentration of empagliflozin in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa/1000 mg Glumetza® (Fasted) | Empa/ 1000 mg Met FDC (Fasted) | Empa/1000 mg Glumetza ® (Fed) | Empa/ 1000 mg Met FDC (Fed) | Empa/ 1500 mg Glumetza® (Fasted) | Empa/ 1500 mg Met FDC (Fasted)
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 24 | 23
nmol/L | 377 (22.5) | 395 (24.6) | 273 (27.6) | 277 (31.0) | 396 (21.9) | 381 (22.0)
Statistical Analysis 1: Comparison: Empa/1000 mg Glumetza® (Fasted) vs Empa/ 1000 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 104.83, 90% CI 2-sided [99.522 to 110.412], Standard Error of Mean 1.031 — Ratio calculated as Empa/ 1000 mg Met FDC (Fasted) divided by Empa/1000 mg Glumetza® (Fasted)
Statistical Analysis 2: Comparison: Empa/1000 mg Glumetza ® (Fed) vs Empa/ 1000 mg Met FDC (Fed); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 101.84, 90% CI 2-sided [95.030 to 109.134], Standard Error of Mean 1.041 — Ratio calculated as Empa/ 1000 mg Met FDC (Fed) divided by Empa/1000 mg Glumetza ® (Fed)
Statistical Analysis 3: Comparison: Empa/ 1500 mg Glumetza® (Fasted) vs Empa/ 1500 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 96.03, 90% CI 2-sided [90.217 to 102.211], Standard Error of Mean 1.037 — Ratio calculated as Empa/ 1500 mg Met FDC (Fasted) divided by Empa/ 1500 mg Glumetza® (Fasted)

5. Primary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma, for Metformin
Description: Maximum measured concentration of metformin in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Empa/1000 mg Glumetza® (Fasted) | Empa/ 1000 mg Met FDC (Fasted) | Empa/1000 mg Glumetza ® (Fed) | Empa/ 1000 mg Met FDC (Fed) | Empa/ 1500 mg Glumetza® (Fasted) | Empa/ 1500 mg Met FDC (Fasted)
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 24 | 23
ng/mL | 975 (37.2) | 964 (39.9) | 1110 (21.2) | 1200 (22.7) | 1220 (32.8) | 1270 (34.7)
Statistical Analysis 1: Comparison: Empa/1000 mg Glumetza® (Fasted) vs Empa/ 1000 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p = 0.0027, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 98.94, 90% CI 2-sided [87.925 to 111.329], Standard Deviation 1.071 — Ratio calculated as Empa/ 1000 mg Met FDC (Fasted) divided by Empa/1000 mg Glumetza® (Fasted)
Statistical Analysis 2: Comparison: Empa/1000 mg Glumetza ® (Fed) vs Empa/ 1000 mg Met FDC (Fed); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 108.18, 90% CI 2-sided [102.792 to 113.859], Standard Error of Mean 1.030 — Ratio calculated as Empa/ 1000 mg Met FDC (Fed) divided by Empa/1000 mg Glumetza ® (Fed)
Statistical Analysis 3: Comparison: Empa/ 1500 mg Glumetza® (Fasted) vs Empa/ 1500 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p = 0.0060, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 103.62, 90% CI 2-sided [92.116 to 116.559], Standard Error of Mean 1.071 — Ratio calculated as Empa/ 1500 mg Met FDC (Fasted) divided by Empa/ 1500 mg Glumetza® (Fasted)

6. Secondary Outcome: AUC0-infinity (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity), for Metformin
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Empa/1000 mg Glumetza® (Fasted) | Empa/ 1000 mg Met FDC (Fasted) | Empa/1000 mg Glumetza ® (Fed) | Empa/ 1000 mg Met FDC (Fed) | Empa/ 1500 mg Glumetza® (Fasted) | Empa/ 1500 mg Met FDC (Fasted)
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 24 | 23
ng*h/mL | 7480 (37.4) | 7360 (36.7) | 13900 (20.7) | 13600 (20.4) | 10500 (28.5) | 10900 (28.7)
Statistical Analysis 1: Comparison: Empa/1000 mg Glumetza® (Fasted) vs Empa/ 1000 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p = 0.0008, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 98.33, 90% CI 2-sided [89.13 to 108.47], Standard Error of Mean 1.06 — Ratio calculated as Empa/ 1000 mg Met FDC (Fasted) divided by Empa/1000 mg Glumetza® (Fasted)
Statistical Analysis 2: Comparison: Empa/1000 mg Glumetza ® (Fed) vs Empa/ 1000 mg Met FDC (Fed); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p < 0.0001, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 98.71, 90% CI 2-sided [94.77 to 102.80], Standard Error of Mean 1.02 — Ratio calculated as Empa/ 1000 mg Met FDC (Fed) divided by Empa/1000 mg Glumetza ® (Fed)
Statistical Analysis 3: Comparison: Empa/ 1500 mg Glumetza® (Fasted) vs Empa/ 1500 mg Met FDC (Fasted); Test type: Non-Inferiority or Equivalence — Model includes effects for sequence, subjects within sequences, period and treatment; p = 0.0021, ANOVA; P-value for ratio outside interval 80%-125%; Adjusted geometric mean ratio (%) = 103.90, 90% CI 2-sided [94.09 to 114.74], Standard Error of Mean 1.06 — Ratio calculated as Empa/ 1500 mg Met FDC (Fasted) divided by Empa/ 1500 mg Glumetza® (Fasted)

ADVERSE EVENTS:
Time Frame: From drug administration until next treatment period or follow-up visit, 10 days
Arm/Group | Empa/1000 mg Glumetza® (Fasted) | Empa/ 1000 mg Met FDC (Fasted) | Empa/1000 mg Glumetza ® (Fed) | Empa/ 1000 mg Met FDC (Fed) | Empa/ 1500 mg Glumetza® (Fasted) | Empa/ 1500 mg Met FDC (Fasted)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 4/24 | 5/24 | 4/24 | 4/24 | 6/24 | 7/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa/1000 mg Glumetza® (Fasted) (N=24) | Empa/ 1000 mg Met FDC (Fasted) (N=24) | Empa/1000 mg Glumetza ® (Fed) (N=24) | Empa/ 1000 mg Met FDC (Fed) (N=24) | Empa/ 1500 mg Glumetza® (Fasted) (N=24) | Empa/ 1500 mg Met FDC (Fasted) (N=23)
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 1 | 4 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.